CLINICAL TRIAL: NCT00809016
Title: Contribution of Positron Emission Tomography in Biological Targeting by Conformational Radiotherapy and Intensity-modulated Radiotherapy of Ear, Nose and Throat Tumors
Brief Title: PET Scans in Patients With Head And Neck Cancer Who Are Undergoing 3-Dimensional Conformal Radiation Therapy And Intensity-Modulated Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000626776; COL-0606; COL-TEPORL; COL-RCB 2007-A00291-52; INCA-RECF0488
Record Dates: First submitted 2008-12-13; First posted 2008-12-16 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2009-07

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV squamous cell carcinoma of the lip and oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Radiotherapy, Conformal; Fluorodeoxyglucose F18; Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy
Radiation: fludeoxyglucose F 18
Radiation: intensity-modulated radiation therapy

SUMMARY:
RATIONALE: Imaging procedures, such as PET scans, may determine the extent of cancer and help doctors plan radiation therapy. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy that uses a 3-dimensional image of the tumor to help focus thin beams of radiation directly on the tumor, and giving radiation therapy in higher doses over a shorter period of time, may kill more tumor cells and have fewer side effects. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This clinical trial is studying PET scans to see how well they work in patients with head and neck cancer who are undergoing 3-dimensional conformal radiation therapy and intensity-modulated radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the value of pre-treatment PET in determining the target volume in patients with head and neck cancer undergoing three-dimensional conformational radiotherapy and intensity-modulated radiotherapy.

Secondary

* To evaluate variations in weekly fludeoxyglucose F 18 PET imaging during the first 5 weeks of treatment.
* To determine the relationship between changes in tumor metabolism during radiotherapy and control tumor at 3 months and at 1 year post-treatment.

OUTLINE: This is a multicenter study.

Patients undergo fludeoxyglucose F18 PET (FDG-PET) in addition to conventional imaging at baseline. Patients undergo standard three-dimensional conformational radiotherapy and intensity-modulated radiation therapy 5 days a week for 5 weeks.

Some patients also undergo weekly FDG-PET during treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed head and neck cancer

  * No nasopharyngeal or paranasal sinus cancer
  * Locally advanced disease (T3 or T4)
  * Not in complete remission
* Planning to undergo curative radiotherapy (minimum dose of 66 Gy), with or without standard treatment (i.e., platinum-based chemotherapy or biological therapy/rituximab)
* Measurable tumor according to RECIST criteria

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Not pregnant or nursing
* Able to lie still for 1 hour
* No history of progressive neoplastic disease
* No known hypersensitivity to fludeoxyglucose F18 or any of its excipients
* No severe or uncontrolled systemic disease, including any of the following:

  * Kidney disease
  * Liver disease
  * Cardiac disease
  * Unstable or uncompensated respiration
  * Uncontrolled diabetes (i.e., glucose ≥ 1.5 g/L)
* No geographical, social, or psychological conditions that make follow-up impossible

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior surgery
* No concurrent experimental agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-05; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Difference between the target volume to be irradiated as measured by conventional imagining and PET

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lartigau, MD, PhD — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, France